CLINICAL TRIAL: NCT05646693
Title: Effect of Combined Antioxidant Therapy on Oxidative Stress Markers and Inflammatory in Patients With Chronic Subjective Endotic Tinnitus
Brief Title: Effect of Combined Antioxidant Therapy on Oxidative Stress Markers and Inflammatory Cytokines in Patients With Tinnitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Institute of Experimental and Clinical Therapeutics (Unknown); Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Adolfo Daniel Rodriguez-Carrizalez, Research Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACSE202208/IIA
Record Dates: First submitted 2022-11-25; First posted 2022-12-12 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Tinnitus, Subjective; Tinnitus, Bilateral; Antioxidant Therapy; Psychiatric Drugs; Oxidative Stress; Inflammatory Cytokines; SSRI
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Geritol; Sertraline; Magnesium Oxide

STUDY DESIGN:
Intervention Model Description: Clinical Trial Phase II A, controlled with placebo
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drusen Mega® + Sertraline (Experimental): It will consist of 29 patients with Chronic Subjetive Endotic Tinnitus. Patients will eat one capsule of antioxidant therapy (Drusen Mega®) and one capsule of sertraline per day in the night for 3 months.
  Interventions: Dietary Supplement: Drusen Mega®; Drug: Sertraline
- Placebo + Sertraline (Placebo Comparator): It will consist of 29 patients with Chronic Subjetive Endotic Tinnitus. Patients will eat one capsule of placebo (Magnesium Oxide 100mg) per day in the morning and one capsule of sertraline per day in the night for 3 months.
  Interventions: Drug: Sertraline; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Drusen Mega® — It consists of a dietary supplement composed of Vitamin C 60.0mg, Vitamin E 30.0mg, Zinc 12.5mg, Copper 1.0mg, Astaxanthin 4.0mg, Zeaxanthin 2.0mg, Lutein 10.0mg and Omega 3 Acids 500.0mg. It is suggested to consume one capsule per day, preferably with food. This supplement is indicated for nutritional deficiencies and in patients with ophthalmological pathologies.
  Other Names: Multivitamins
  Arms: Drusen Mega® + Sertraline
Drug: Sertraline — It consists of a drug capsule composed of Sertraline Hydrochloride 50mg. In adults it is suggested to consume one to four capsule(s) per day, administering (preferably) the highest dose in the evening, before going to bed. This drug is indicated in the treatment of depressive states with anxiety or moderate to severe agitation, which are accompanied by tension, excitement, insomnia, obsessive and hypochondriac traits. It is also indicated in obsessive-compulsive disorder, panic attacks, stress disorder, post-traumatic disorder, social anxiety disorder and used to relieve the symptoms of premenstrual dysphoric disorder.
  Other Names: Sertraline Hydrochloride
Drug: Placebo — It consists of a placebo capsule composed of Magnesium Oxide 100mg. This component is inert in the dose at which it will be administered.
  Other Names: Magnesium Oxide
  Arms: Placebo + Sertraline

SUMMARY:
The main objective of our study is to evaluate the effect of combinated antioxidants therapy with Adepsique® (amitriptyline, perphenazine, and diazepam) on patients with tinnitus chronic symptoms, evaluating the levels of inflammatory cytokines and oxidative stress in blood.

The researchers intend to include 58 patients, divided into two intervention groups, who will be randomly assigned a pill with antioxidants or placebo, and the patient must eat one pill per day for 3 months.

In the study, the clinical characteristics of tinnitus, inflammatory cytokines and oxidative stress markers will be evaluated, before, during and after the intervention with antioxidant therapy. Subsequently, the clinical and sample results will be evaluated to compare the effects between them.

DETAILED DESCRIPTION:
Tinnitus is a pathology defined as the perception of a sound without an external acoustic stimulus. About 15 to 20% of the world population suffers from this pathology.It is classified according to the time of presentation (acute or chronic); in the existence of an internal source measurable and perceptible by the patient and the physician (objective) or where the source does not exist and is only perceived by the patient (subjective), the latter being the most common. And, in the place where they originate, exotic (outside the ear), endotic (within the auditory apparatus), and central (within the cerebral cortex without lesion of the auditory apparatus). As well as the influence it presents in daily life, being mild, moderate, severe or catastrophic.

Within the pathophysiology, the influence of different proinflammatory cytokines such as IL-6, TNF-α, β-2GP1, IL-1, among others, is described; as well as markers of oxidative stress and elevated levels of ROS, which annul defense mechanisms against oxidative damage, and induce damage to DNA, lipids, and membrane proteins.ncreased levels of nitric oxide, peroxynitrite, nuclear transcriptional factor Kappa-B (NF-κB), glutamate (N-methyl D-aspartate) receptors, and calcium cause hair cell damage. On the other hand, reduced levels of antioxidant enzymes such as superoxide dismutase, glutathione peroxidase, glutathione reductase, catalase, and glutathione transferase perpetuate cell damage.

The diagnosis is based mainly on ruling out etiological factors, associated symptoms or existing comorbidities that cause tinnitus secondarily, as well as a detailed clinical history, measurement of hearing quality, and demonstration of the imbalance of neurotransmitters and proinflammatory molecules.

Because it is a multifactorial entity, the definitive treatment has not yet been developed. Extensive pharmacological therapies, from the use of NSAIDs to antidepressant and antipsychotic drugs, have been tried with ambiguous, inconsistent and inconclusive results. Alternative therapies with multivitamins and antioxidants have shown probable utility in the treatment of tinnitus, however, the existing evidence is of poor and conflicting quality.The latter reduce oxidative stress through different means; through the destruction of free radicals by donating electrons to the unpaired states of these radicals. Another means is through the catalysis of free radicals, converting them into harmless molecules (water and oxygen). Lastly, they support reducing chronic inflammation secondarily by decreasing the rate of auditory hairy cell apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with subjective chronic tinnitus (unilateral or bilateral)
* Patients with normal audiometry or identification of hearing loss up to a medium degree (20-70 dB)
* Patients with evidence of endotic tinnitus
* Patients who have or do not have social medical security
* Females of childbearing age with a negative pregnancy test and use of oral contraceptives
* Patients under pharmacological management with a period of stable medication (≥3 months) for chronic degenerative diseases and under good metabolic control (according to ADA 2022 criteria) through primary intervention

Exclusion Criteria:

* Presence of tinnitus secondary to head trauma, acoustic trauma, or sudden hearing loss
* History or presence of Ménière's disease, otosclerosis, acute or chronic otitis media
* Active gastrointestinal haemorrhagic disease
* History or presence of cancer (any type) or submission to radio and/or chemotherapy
* Autoimmune disease (any)
* History of severe cardiovascular disease (myocardial infarction, stroke, severe peripheral vascular disease)
* Benign prostatic hyperplasia
* Blood dyscrasias and/or bleeding diathesis
* Thyroid disease (any)
* Temporomandibular joint dysfunction
* Neurodegenerative processes
* Hepatic and renal failure
* Closed or open angle glaucoma
* Intake of any medication belonging to the following families (Anticoagulants, Benzodiazepines, ASA diuretics, Aminoglycosides, Chemotherapeutics, Acetylsalicylic Acid, Quinine, MAOIs)
* Intake of antioxidants in the last 6 months
* Hypersensitivity to vitamins that constitute the antioxidant intervention, or any medication belonging to the Adepsique formulation
* Pregnancy, lactation
* History of disease due to COVID-19 infection in the last 6 months
* Diet rich in antioxidants that exceeds the concentrations of the daily nutritional recommendations of the Dietary Reference Intake
* Participation in another clinical trial
* Drug abuse, smoking (daily consumption during the last month of 5 to 10 cigarettes) and/or alcoholism

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in levels of Superoxide Dismutase (SOD) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The enzyme concentration will be determined with multiplex bead immunoassays technique and reported in microunits per milliliter units (mUI/mL)
Change from baseline in levels of Catalase (CAT) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The enzyme concentration will be determined with multiplex bead immunoassays technique and reported in microunits per milliliter units (mUI/mL)
Change from baseline in levels of Glutathione Peroxidase (GPx) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The enzyme concentration will be determined with multiplex bead immunoassays technique and reported in microunits per milliliter units (mUI/mL)
Change from baseline in levels of Malondialdehyde (MDA) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The enzyme concentration will be determined with multiplex bead immunoassays technique and reported in microunits per milliliter units (mUI/mL)
Change from baseline in levels of Oxidized Low-Density Lipoprotein LDL (oxLDL) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The enzyme concentration will be determined with multiplex bead immunoassays technique and reported in nanograms per milliliter units (ng/mL)
Change from baseline in levels of Tumor Necrosis Factor Alpha (TNF-a) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of Interleukin 8 (IL-8) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of Interleukin 6 (IL-6) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of Gamma Interferon (IFN-γ) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of Nuclear Factor Kappa B (NF-κB) | 90 days
  Standard blood sampling will be collected through a catheter in an antecubital vein in tubes without EDTA, centrifuged and serum will placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in nanogram per milliliter units (ng/mL)

SECONDARY OUTCOMES:
Change from baseline in Tinnitus Loudness (db) Assessment | 90 days
  Tinnitus screening tests will be conducted, using psychoacoustic techniques including pitch loudness matching within a soundproof booth. Patients will be given pairs of different tones in the non-tinnitus or less intense ear and will be asked to choose which tone is closest to the perceived tinnitus. This will be continued until a definite match will made. The results will be expressed in decibels
Change from baseline in Tinnitus Frecuency (Hz) Assessment | 90 days
  Tinnitus screening tests will be conducted, using psychoacoustic techniques including pitch frequency matching within a soundproof booth. Patients will be given pairs of different tones in the non-tinnitus or less intense ear and will be asked to choose which tone is closest to the perceived tinnitus. This will be continued until a definite match will made. The results will be expressed in hertz.
Change from baseline in Audiometric Assessment | 90 days
  Patients will undergo conventional pure tone audiometry and extended high frequency (EHF) audiometry to determine any hearing loss. The degree of hearing loss will be determined using the average of values in four consecutive frequencies (500-1000-2000-4000) and will be classified as normal hearing, little, mild, moderate or severe hearing loss.
Change from baseline in Tinnitus Discomfort Assessment | 90 days
  Patients will complete the questionnaire Tinnitus Handicap Inventory (THI) which measure the subjective discomfort a patient experiences because of tinnitus. THI comprises 25 questions which are divided in functional, emotional, and catastrophic subscales. Total scores of THI range from 0 to 100.
Change from baseline in levels of Otolin-1 | 90 days
  Otolin-1 is a scaffold glycoprotein that connects the otoliths and matrix proteins of the otoconial nucleus with the sensory epithelium. Under normal conditions it is not found in peripheral blood, but in some hearing diseases it can be measured due to the loss of the blood-cochlear barrier. This will serve as an ear-specific marker.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo D Rodríguez-Carrizalez, MD / PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics,, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be shared. The data is protected under the Mexican Federal Law for the Protection of Personal Data Held by Private Parties.

REFERENCES:
- [Background] Henry JA, Dennis KC, Schechter MA. General review of tinnitus: prevalence, mechanisms, effects, and management. J Speech Lang Hear Res. 2005 Oct;48(5):1204-35. doi: 10.1044/1092-4388(2005/084). PMID 16411806
- [Background] Weber C, Arck P, Mazurek B, Klapp BF. Impact of a relaxation training on psychometric and immunologic parameters in tinnitus sufferers. J Psychosom Res. 2002 Jan;52(1):29-33. doi: 10.1016/s0022-3999(01)00281-1. PMID 11801262
- [Background] Gomaa NA, Jimoh Z, Campbell S, Zenke JK, Szczepek AJ. Biomarkers for Inner Ear Disorders: Scoping Review on the Role of Biomarkers in Hearing and Balance Disorders. Diagnostics (Basel). 2020 Dec 29;11(1):42. doi: 10.3390/diagnostics11010042. PMID 33383894
- [Background] Solis-Angeles S, Juarez-Perez CA, Jimenez-Ramirez C, Cabello-Lopez A, Aguilar-Madrid G, Del Razo LM. Prestin and otolin-1 proteins in the hearing loss of adults chronically exposed to lead. Toxicol Appl Pharmacol. 2021 Sep 1;426:115651. doi: 10.1016/j.taap.2021.115651. Epub 2021 Jul 15. PMID 34273409
- [Background] Esmaili AA, Renton J. A review of tinnitus. Aust J Gen Pract. 2018 Apr;47(4):205-208. doi: 10.31128/AJGP-12-17-4420. PMID 29621860
- [Background] Celik M, Koyuncu I. A Comprehensive Study of Oxidative Stress in Tinnitus Patients. Indian J Otolaryngol Head Neck Surg. 2018 Dec;70(4):521-526. doi: 10.1007/s12070-018-1464-7. Epub 2018 Jul 27. PMID 30464909
- [Background] Polanski JF, Soares AD, de Mendonca Cruz OL. Antioxidant therapy in the elderly with tinnitus. Braz J Otorhinolaryngol. 2016 May-Jun;82(3):269-74. doi: 10.1016/j.bjorl.2015.04.016. Epub 2015 Oct 17. PMID 26547700
- [Background] Pawlak-Osinska K, Kazmierczak H, Marzec M, Kupczyk D, Bilski R, Mikolajewska E, Mikolajewski D, Augustynska B. Assessment of the State of the Natural Antioxidant Barrier of a Body in Patients Complaining about the Presence of Tinnitus. Oxid Med Cell Longev. 2018 Oct 28;2018:1439575. doi: 10.1155/2018/1439575. eCollection 2018. PMID 30510615
- [Background] Petridou AI, Zagora ET, Petridis P, Korres GS, Gazouli M, Xenelis I, Kyrodimos E, Kontothanasi G, Kaliora AC. The Effect of Antioxidant Supplementation in Patients with Tinnitus and Normal Hearing or Hearing Loss: A Randomized, Double-Blind, Placebo Controlled Trial. Nutrients. 2019 Dec 12;11(12):3037. doi: 10.3390/nu11123037. PMID 31842394
- [Result] Baguley D, McFerran D, Hall D. Tinnitus. Lancet. 2013 Nov 9;382(9904):1600-7. doi: 10.1016/S0140-6736(13)60142-7. Epub 2013 Jul 2. PMID 23827090